CLINICAL TRIAL: NCT02708212
Title: Optimal Procedural Sequence in Same-day Bidirectional Endoscopy With Moderate Sedation and Carbon Dioxide Insufflation: A Prospective Randomized Controlled Study
Brief Title: Optimal Procedural Sequence in Same-day Bidirectional Endoscopy: A Prospective Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evergreen General Hospital, Taiwan (Other)
Responsible Party: Principal Investigator, Chi-Liang Cheng, M.D., Evergreen General Hospital, Taiwan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: ZEH-2016-2
Record Dates: First submitted 2016-03-06; First posted 2016-03-15 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Endoscopy; Moderate Sedation
MeSH Terms: interventions — Endoscopy, Digestive System; Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGD-colonoscopy group (Active Comparator): In this group, patients receiving an EGD followed by a colonoscopy during a same-day bidirectional endoscopy. Patients receive moderate conscious sedation with fentanyl and midazolam for the procedures. Gastric polypectomy will be provided when gastric polyps are found during an EGD study. Colon polypectomy will be provided when colon polyps are found during a colonoscopy study. Patients' heart rate, respiratory rate, blood pressure, and oxygen saturation will be recorded every 60 seconds during the endoscopic examinations. Patients' tolerability to EGD and colonoscopy examinations will be scaled by patients and endoscopists after the completion of the examinations. Aldrete scores are recorded15 minutes and 25 minutes after entering the recovery room. The recovery time will also be recorded.
  Interventions: Procedure: EGD and colonoscopy
- Colonoscopy-EGD group (Active Comparator): In this study group, patients receive a colonoscopy followed by an EGD during a same-day bidirectional endoscopy. Patients receive moderate conscious sedation with fentanyl and midazolam for the procedures. Colon polypectomy will be provided when colon polyps are found during a colonoscopy study. Gastric polypectomy will be provided when gastric polyps are found during an EGD study. Patients' heart rate, respiratory rate, blood pressure, and oxygen saturation will be recorded every 60 seconds during the endoscopic examinations. Patients' tolerability to colonoscopy and EGD examinations will be scaled by patients and endoscopists after the completion of the examinations. Aldrete scores are recorded15 minutes and 25 minutes after entering the recovery room. The recovery time will also be recorded.
  Interventions: Procedure: EGD and colonoscopy

INTERVENTIONS:
Procedure: EGD and colonoscopy — Cold forceps biopsy, cold snare polypectomy, and/or hot snare polypectomy will be performed for stomach and/or colon polyps during EGD and colonoscopy examinations will be performed whenever indicated.

SUMMARY:
The Same-day bidirectional endoscopy (BDE) is commonly used in clinical practice. However, the optimal sequence of performing a same-day BDE has not been well-established.The primary aims of this study are to compare the sedative doses and patient discomfort between the study groups who received a colonoscopy followed by and EGD (colonoscopy-EGD), or an EGD followed by a colonoscopy (EGD-colonoscopy) during a same-day BDE. The secondary aim is to assess colonoscopy performance, including the cecal intubation time and adenoma detection rate between the two endoscopic sequences.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, aged 20 to 75 years, who are scheduled for same-day bidirectional endoscopy examination for any indication are invited to participate in the study.

Exclusion Criteria:

* 1. previous gastrectomy or colectomy 2. inadequate bowel preparation, 3. obstructive lesions of the colon 4. severe colitis, gastrointestinal bleeding 5. allergy to fentanyl or midazolam 6. American Society of Anesthesiology (ASA) classification of physical status grade 3 or higher, 7. mental retardation 8. regular use of narcotics 9. pregnancy 10. refusal to provide a written informed consent.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Liang Cheng, MD, Principal Investigator — Evergreen General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 129 patients were invited to participate in the study from April to July 2016, and 8 patients were excluded. Finally, 121 patients were recruited for the study which was performed in a community hospital (Evergreen General Hospital). One patient in the EGD-colonoscopy was further excluded from final analysis due to poor bowel preparation.
Pre-assignment Details: Eight patients were excluded from assignment due to refusal to provide informed consent (n=3), American Society of Anesthesiology class 3 (n=3), duodenal peptic stricture (n =1), and partial colectomy (n=1).
Groups:
- EGD-colonoscopy Group: In this study group, 60 patients received an EGD followed by a colonoscopy during a same-day bidirectional endoscopy. Patients received modeate conscious sedation with fentanyl and midazolam and carbon dioxide insullfation. Interventions with cold forceps polypectomy, cold snare polypectomy or hot snare polypectomy were performed for gastric and/or colon polyps during endoscopy procedures. Patients' heart rate, respiratory rate, blood pressure, and oxygen saturation were recorded every 60 seconds during endoscopic examinations. Patients' tolerability to both endoscopy examinations was scaled by patients and endoscopists after examinations. Aldrete scores, at 15 minutes and 25 minutes after entering the recovery room, was recorded. Recovery time to discharge was also recorded.
- Colonoscopy-EGD Group: In this study group, 60 patients received a colonoscopy followed by and an EGD during a same-day bidirectional endoscopy. Patients received modeate conscious sedation with fentanyl and midazolam and carbon dioxide insufflation. Interventions with cold forceps polypectomy, cold snare polypectomy or hot snare polypectomy were performed for gastric and/or colon polyps during EGD and colonoscopy examinations. Patients' heart rate, respiratory rate, blood pressure, and oxygen saturation were recorded every 60 seconds during endoscopic examinations. Patients' tolerability to both endoscopy examinations was scaled by patients and endoscopists after examinations. Aldrete scores, at 15 minutes and 25 minutes after entering the recovery room, were recorded. Recovery time to discharge was also recorded.
Period: Overall Study
Arm/Group | EGD-colonoscopy Group | Colonoscopy-EGD Group
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total 120 patients were randomly assigned to EGD-colonoscopy group (n=60) and colonoscopy-EGD group (n=60).
Groups:
- EGD-colonoscopy Group: In this study group, 60 patients received an EGD followed by a colonoscopy during a same-day bidirectional endoscopy. Patients received moderate conscious sedation with fentanyl and midazolam and carbon dioxide insufflation. Interventions with cold forceps polypectomy, cold snare polypectomy or hot snare polypectomy were performed for gastric and/or colon polyps during endoscopy procedures. Patients' heart rate, respiratory rate, blood pressure, and oxygen saturation were recorded every 60 seconds during endoscopic examinations. Patients' tolerability to both endoscopy examinations was scaled by patients and endoscopists after examinations. Aldrete scores, at 15 minutes and 25 minutes after entering the recovery room, was recorded. Recovery time to discharge was also recorded.
- Colonoscopy-EGD Group: In this study group, 60 patients received a colonoscopy followed by and an EGD during a same-day bidirectional endoscopy. Patients received moderate conscious sedation with fentanyl and midazolam and carbon dioxide insufflation. Interventions with cold forceps polypectomy, cold snare polypectomy or hot snare polypectomy were performed for gastric and/or colon polyps during EGD and colonoscopy examinations. Patients' heart rate, respiratory rate, blood pressure, and oxygen saturation were recorded every 60 seconds during endoscopic examinations. Patients' tolerability to both endoscopy examinations was scaled by patients and endoscopists after examinations. Aldrete scores, at 15 minutes and 25 minutes after entering the recovery room, were recorded. Recovery time to discharge was also recorded.
- Total: Total of all reporting groups
Arm/Group | EGD-colonoscopy Group | Colonoscopy-EGD Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.1) | 52.9 (12.7) | 53.7 (11.9)
Gender [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 26 | 30 | 56
Region of Enrollment [Number; unit: participants]
  Taiwan | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Sedative Doses of Fentanyl
Description: During bidirectional endoscopy, the total doses of fentanyl were recorded and compared between the two study groups.
Time Frame: On the day of endoscopic procedures.
Measure: Mean (Standard Deviation); unit: mcg/kg
Groups:
- EGD-colonoscopy Group: In this group, patients received an EGD followed by a colonoscopy during a same-day bidirectional endoscopy. Moderate conscious sedation with fentanyl and midazolam was provided. The total doses of fentanyl after the completion of bidirectional endoscopy were recorded.
  EGD and colonoscopy: Gastric polypectomy was provided when gastric polyps were found during an EGD study. Colon polypectomy was provided when colon polyps were found during a colonoscopy study.
- Colonoscopy-EGD Group: In this group, patients received a colonoscopy followed by an EGD during a same-day bidirectional endoscopy. Moderate conscious sedation with fentanyl and midazolam was provided. The total doses of fentanyl after the completion of bidirectional endoscopy were recorded.
  EGD and colonoscopy: Gastric polypectomy was provided when gastric polyps were found during an EGD study. Colon polypectomy was provided when colon polyps were found during a colonoscopy study.
Arm/Group | EGD-colonoscopy Group | Colonoscopy-EGD Group
Number analyzed (Participants) | 60 | 60
mcg/kg | 1.09 (0.42) | 1.28 (0.31)
Statistical Analysis 1: Comparison: EGD-colonoscopy Group vs Colonoscopy-EGD Group; The two-sample t test will be used to compare the total doses of fentanyl and midazolam between the two study groups; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Sedative Doses of Midazolam
Description: During bidirectional endoscopy, the total doses of midazolam were recorded and compared between the two study groups.
Time Frame: On the day of bidirectional endoscopy procedures
Measure: Mean (Standard Deviation); unit: mg/kg
Groups:
- EGD-colonoscopy Group: In this group, patients received an EGD followed by a colonoscopy during a same-day bidirectional endoscopy. Moderate conscious sedation with fentanyl and midazolam was provided. The total doses of midazolam after the completion of the bidirectional endoscopy were recorded.
  EGD and colonoscopy: Gastric polypectomy was provided when gastric polyps were found during an EGD study. Colon polypectomy was provided when colon polyps were found during a colonoscopy study.
- Colonoscopy-EGD Group: In this group, patients received a colonoscopy followed by an EGD during a same-day bidirectional endoscopy. Moderate conscious sedation with fentanyl and midazolam was provided. The total doses of midazolam after the completion of the bidirectional endoscopy were recorded.
  EGD and colonoscopy: Gastric polypectomy was provided when gastric polyps were found during an EGD study. Colon polypectomy was provided when colon polyps were found during a colonoscopy study.
Arm/Group | EGD-colonoscopy Group | Colonoscopy-EGD Group
Number analyzed (Participants) | 60 | 60
mg/kg | 0.08 (0.03) | 0.10 (0.02)
Statistical Analysis 1: Comparison: EGD-colonoscopy Group; The two-sample t test will be used to compare the total doses of midazolam between the two study groups; Test type: Superiority or Other; p = 0.0012, t-test, 2 sided

3. Secondary Outcome: Overall Duration of BDE Examinations
Description: The overall duration of both EGD and colonoscopy examinations was recorded and compared.
Time Frame: On the day of bidirectional endoscopy
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- EGD-colonoscopy Group: The duration of both EGD and colonoscopy examinations was recorded and compared.
- Colonoscopy-EGD Group: The duration of both colonoscopy and EGD examinations was recorded and compared.
Arm/Group | EGD-colonoscopy Group | Colonoscopy-EGD Group
Number analyzed (Participants) | 60 | 60
minutes | 32.7 (9.9) | 33.3 (7.5)
Statistical Analysis 1: Comparison: EGD-colonoscopy Group vs Colonoscopy-EGD Group; Test type: Superiority or Other; p = 0.6967, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the start of bidirectional endoscopy to one hour after the completion of the bidirectional endoscopy.
Description: The adverse events during moderate sedation were usually transient and related to overall sedative doses. The primary aim of the study was to compared the overall sedative doses between the patients receiving EGD-colonoscopy and colonoscopy-EGD sequences. Theoretically, patients who received less sedative doses should experience less episodes of adverse events. Therefore, we calculated the overall sedative doses and adverse events after the completion of both EGD and colonoscopy examinations.
Groups:
- EGD-colonoscopy Group; Colonoscopy-EGD Group: Patients received moderate conscious sedation with fentanyl and midazolam. Blood pressure, heart rate, and oxygen saturation were monitored and recorded during the endoscopic procedures. Supplemental oxygen (2 L/min) by nasal cannula was provided for every patient. The following adverse events were recorded during conscious sedation: 1) oxygen desaturation: < 90% persisting for more than 60 s; 2) hypotension: < 90 mm Hg systolic blood pressure for more than 60 s; 3) hypertension: > 180 mm Hg systolic blood pressure for more than 60 s; 4) tachycardia: > 120 beats per minute, lasting more than 60 s; and 5) bradycardia: < 50 beats per minute, lasting more than 60 s.
Arm/Group | EGD-colonoscopy Group | Colonoscopy-EGD Group
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 19/60 | 20/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGD-colonoscopy Group (N=60) | Colonoscopy-EGD Group (N=60)
Transient hypotension (Vascular disorders) | 19 (19) | 20 (20) — 20 patients (33.3%) in the colonoscopy-EGD group and 19 patients (31.7%) in the EGD-colonoscopy group developed transient hypotension during the bidirectional endoscopy examinations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No